CLINICAL TRIAL: NCT01616004
Title: Effect of Acute Treatment With N2O on Inhibitory Pain Mechanisms in Healthy Subject
Acronym: N2O
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TASMC-12-SB-340-CTIL
Record Dates: First submitted 2012-06-03; First posted 2012-06-11 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Nitrous Oxide; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N2O (Experimental): N20 70% inhalation 5 minutes O2 100 % inhalation for 5 minutes
  Interventions: Drug: N2O
- Air (Sham Comparator)
  Interventions: Drug: Air

INTERVENTIONS:
Drug: N2O
  Other Names: laughing gas
  Arms: N2O
Drug: Air — sham comparator
  Arms: Air

SUMMARY:
The purpose of this study is to determine whether N2O (laughing gas) has an antinociceptive effects in healthy volunteers.

DETAILED DESCRIPTION:
10 healthy volunteers will come twice to the pain medicine unit, at 1 visit they'll get N2O and in the second visit they'll get air as placebo, they won't know what they're getting. During the visit they'll get heat stimulus using QST and will have to report their pain using eVAS (scale from 0 to 100 when 0 is no pain and 100 is the worst pain imagine).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* women and men
* healthy

Exclusion Criteria:

* smokers
* medication use pregnant woman cardiovascular disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | August 2016

CONTACTS AND LOCATIONS:
Overall Officials: Silviu Brill, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel